CLINICAL TRIAL: NCT00096018
Title: A Phase I/II Study of Fludarabine Plus Thalidomide as Frontline Therapy for Newly Diagnosed Patients With Chronic Lymphocytic Leukemia
Brief Title: Fludarabine and Thalidomide in Treating Patients With Newly Diagnosed Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000391769; RPC-01-12
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Results first posted 2013-03-05 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-09

CONDITIONS: Leukemia
Keywords: stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine phosphate; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose escalation (Experimental): Thalidomide (100 mg/day, 200 mg/day, or 300 mg/day) on Day 1 followed by Fludarabine 25 mg/m2/day for 5 days starting on Day 7 (cycle = 28 days
  Interventions: Drug: fludarabine phosphate; Drug: thalidomide

INTERVENTIONS:
Drug: fludarabine phosphate — Given IV
Drug: thalidomide — Orally

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine, work in different ways to stop cancer cells from dividing so they stop growing or die. Biological therapies such as thalidomide use different ways to stimulate the immune system and stop cancer cells from growing. Combining fludarabine with thalidomide may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of thalidomide when given together with fludarabine and to see how well they work in treating patients with newly diagnosed B-cell chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and efficacy of fludarabine and thalidomide in patients with newly diagnosed B-cell chronic lymphocytic leukemia.
* Determine the overall response rate (complete and partial) in patients treated with this regimen.
* Determine the duration of response in patients treated with this regimen.

OUTLINE: This is an open-label, phase I, dose-escalation study of thalidomide followed by a phase II study.

* Phase I: Beginning on day 1, patients receive oral thalidomide once daily for up to 6 months. Beginning on day 7, patients also receive fludarabine IV over 30 minutes daily for 5 days. Treatment with fludarabine repeats every 28-35 days for up to 6 courses. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of thalidomide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive fludarabine and thalidomide as in phase I at the MTD.

Patients are followed at 4 weeks, every 3 months for 2 years, and then every 4 months for 2 years.

PROJECTED ACCRUAL: Up to 45 patients (≥ 9 for the phase I portion and ≤ 36 for the phase II portion) will be accrued for this study within 8 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of B-cell chronic lymphocytic leukemia (CLL) based on the following criteria:

  * Peripheral blood lymphocytosis > 5,000/mm^3
  * Co-expression of CD5, CD19 or CD20, and CD23 surface antigens
  * Clonal kappa or lambda light chain expression
* No recurrent or refractory CLL
* No other lymphoproliferative diseases or diseases due to transformation of CLL, such as prolymphocytic leukemia or Richter's syndrome

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* At least 12 weeks

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin < 1.5 mg/dL
* AST < 2.5 times upper limit of normal

Renal

* Creatinine ≤ 1.5 mg/dL

Cardiovascular

* No cardiac arrhythmia within the past 6 months
* No myocardial infarction within the past 6 months

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use at least 1 highly active and 1 additional method of contraception for 4 weeks before, during, and for at least 4 weeks after study treatment
* Patients must have sufficient mental capacity to understand the study explanation and provide informed consent
* No other malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix
* No active serious infection uncontrolled by antibiotics
* No medical condition or reason that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No prior therapy for CLL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2002-05; Primary Completion 2010-11 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin Lee, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Result] Chanan-Khan A, Miller KC, Takeshita K, Koryzna A, Donohue K, Bernstein ZP, Mohr A, Klippenstein D, Wallace P, Zeldis JB, Berger C, Czuczman MS. Results of a phase 1 clinical trial of thalidomide in combination with fludarabine as initial therapy for patients with treatment-requiring chronic lymphocytic leukemia (CLL). Blood. 2005 Nov 15;106(10):3348-52. doi: 10.1182/blood-2005-02-0669. Epub 2005 Jul 28. PMID 16051743

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Activated: 3/21/2002. Study Closed: 11/19/2010
Groups:
- Phase I - Dose Escalation: Thalidomide (100 mg/day, 200 mg/day, or 300 mg/day) on Day 1 followed by Fludarabine 25 mg/m2/day for 5 days starting on Day 7 (cycle = 28 days)
- Phase II: Thalidomide 200 mg/day on Day 1 followed by Fludarabine 25 mg/m2/day for 5 days starting on Day 7 (cycle = 28 days)
Period: Overall Study
Arm/Group | Phase I - Dose Escalation | Phase II
Started | 13 | 30
Treated With Study Therapy | 13 | 25
Completed | 11 | 16
Not Completed | 2 | 14
Not completed — Became Ineligible (not treated) | 0 | 3
Not completed — Miscellaneous (not treated) | 0 | 2
Not completed — Adverse Event | 0 | 5
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Miscellaneous | 2 | 1

BASELINE CHARACTERISTICS:
Population: Treated Patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I - Dose Escalation | Phase II | Total
Number analyzed (Participants) | 13 | 25 | 38
Age, Customized [Number; unit: participants]
  30 - 39 years | 2 | 0 | 2
  40 - 49 years | 1 | 2 | 3
  50 - 59 years | 2 | 8 | 10
  60 - 69 years | 5 | 9 | 14
  70 - 79 years | 3 | 6 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 9 | 18 | 27
Region of Enrollment [Number; unit: participants]
  United States | 13 | 25 | 38

OUTCOME MEASURES:

1. Primary Outcome: Overall Responders (Complete and Partial Response)
Description: Criteria for response were based on the Revised National Cancer Institute-sponsored Working Group Guidelines for response, which includes clinical, hematologic, and bone marrow features (Cheson, B.D., et al., National Cancer Institute-sponsored Working Group guidelines for chronic lymphocytic leukemia: revised guidelines for diagnosis and treatment. Blood. 1996;87:4990-97.)
Time Frame: 4 weeks, every 3 months for 2 years, and then every 4 months for 2 years
Population: All Treated Patients
Measure: Number; unit: participants
Arm/Group | Phase I - Dose Escalation | Phase II
Number analyzed (Participants) | 13 | 25
participants | 8 | 18

2. Primary Outcome: Duration of Response
Time Frame: 4 weeks, every 3 months for 2 years, and then every 4 months for 2 years
Population: Patients with Complete or Partial Response
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Phase I - Dose Escalation | Phase II
Number analyzed (Participants) | 8 | 18
months | 43.3 (11.3) | 30.0 (16.4)

ADVERSE EVENTS:
Arm/Group | Phase I - Dose Escalation | Phase II
Serious Adverse Events (participants affected / at risk) | 6/13 | 15/25
Other Adverse Events (participants affected / at risk) | 9/13 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Dose Escalation (N=13) | Phase II (N=25)
Anaemia - Grade 1 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia - Grade 3 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia - Grade 4 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia - Grade 2 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia - Grade 3 (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Febrile neutropenia - Grade 4 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia - Grade 3 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia - Grade 3 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia - Grade 4 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia - Grade 4 (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Angina pectoris - Grade 4 (Cardiac disorders) | 0 (0) | 1 (1)
Death - Grade 5 (General disorders) | 0 (0) | 1 (1)
Fatigue - Grade 2 (General disorders) | 0 (0) | 1 (1)
Fatigue - Grade 3 (General disorders) | 1 (1) | 0 (0)
Oedema peripheral - Grade 1 (General disorders) | 0 (0) | 1 (1)
Pyrexia - Grade 2 (General disorders) | 0 (0) | 1 (1)
Hypersensitivity - Grade 3 (Immune system disorders) | 0 (0) | 1 (1)
Pneumonia - Grade 3 (Infections and infestations) | 0 (0) | 3 (3)
Upper respiratory tract infection - Grade 2 (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection - Grade 3 (Infections and infestations) | 1 (1) | 0 (0)
Femur fracture - Grade 3 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Liver function test abnormal - Grade 4 (Investigations) | 1 (1) | 0 (0)
Decreased appetite - Grade 1 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive - Grade 3 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumour lysis syndrome - Grade 3 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Dysgeusia - Grade 1 (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rash - Grade 3 (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash erythematous - Grade 4 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash generalised - Grade 2 (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Coronary artery bypass - Grade 4 (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis - Grade 3 (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Dose Escalation (N=13) | Phase II (N=25)
Anaemia - Grade 1 (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
Anaemia - Grade 2 (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Anaemia - Grade 3 (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Granulocytopenia - Grade 1 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia - Grade 3 (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Lymphadenopathy - Grade 2 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphopenia - Grade 1 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphopenia - Grade 2 (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymphopenia - Grade 3 (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Neutropenia - Grade 1 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia - Grade 2 (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Neutropenia - Grade 3 (Blood and lymphatic system disorders) | 2 (4) | 5 (7)
Neutropenia - Grade 4 (Blood and lymphatic system disorders) | 2 (3) | 3 (3)
Pancytopenia - Grade 1 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia - Grade 1 (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombocytopenia - Grade 2 (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Thrombocytopenia - Grade 3 (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
Bradycardia - Grade 1 (Cardiac disorders) | 0 (0) | 1 (1)
Ear pain - Grade 1 (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain - Grade 2 (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Diplopia - Grade 2 (Eye disorders) | 0 (0) | 1 (1)
Eye swelling - Grade 1 (Eye disorders) | 0 (0) | 2 (2)
Vision blurred - Grade 1 (Eye disorders) | 0 (0) | 2 (2)
Vision blurred - Grade 2 (Eye disorders) | 0 (0) | 2 (2)
Visual disturbance - Grade 1 (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort - Grade 1 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension - Grade 1 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper - Grade 1 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal tenderness - Grade 1 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation - Grade 1 (Gastrointestinal disorders) | 2 (2) | 5 (5)
Constipation - Grade 2 (Gastrointestinal disorders) | 0 (0) | 4 (4)
Diarrhoea - Grade 1 (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea - Grade 3 (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dry mouth - Grade 1 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia - Grade 1 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence - Grade 1 (Gastrointestinal disorders) | 0 (0) | 1 (2)
Hypoaesthesia oral - Grade 1 (Gastrointestinal disorders) | 0 (0) | 2 (3)
Nausea - Grade 1 (Gastrointestinal disorders) | 2 (2) | 4 (4)
Nausea - Grade 2 (Gastrointestinal disorders) | 0 (0) | 2 (2)
Paraesthesia oral - Grade 1 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting - Grade 1 (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting - Grade 2 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia - Grade 1 (General disorders) | 1 (1) | 4 (4)
Asthenia - Grade 2 (General disorders) | 0 (0) | 2 (2)
Asthenia - Grade 3 (General disorders) | 0 (0) | 1 (1)
Chest pain - Grade 1 (General disorders) | 0 (0) | 1 (1)
Chest pain - Grade 2 (General disorders) | 0 (0) | 1 (1)
Chills - Grade 2 (General disorders) | 0 (0) | 1 (1)
Face oedema - Grade 2 (General disorders) | 0 (0) | 1 (1)
Fatigue - Grade 1 (General disorders) | 2 (2) | 11 (13)
Fatigue - Grade 2 (General disorders) | 1 (1) | 3 (3)
Fatigue - Grade 3 (General disorders) | 0 (0) | 3 (3)
Gait disturbance - Grade 1 (General disorders) | 0 (0) | 1 (1)
Generalised oedema - Grade 1 (General disorders) | 0 (0) | 1 (1)
Influenza like illness - Grade 2 (General disorders) | 0 (0) | 2 (2)
Non-cardiac chest pain - Grade 1 (General disorders) | 0 (0) | 1 (1)
Oedema - Grade 1 (General disorders) | 0 (0) | 1 (1)
Oedema - Grade 2 (General disorders) | 0 (0) | 1 (1)
Oedema peripheral - Grade 1 (General disorders) | 2 (2) | 7 (8)
Oedema peripheral - Grade 2 (General disorders) | 1 (1) | 2 (2)
Pain - Grade 1 (General disorders) | 0 (0) | 2 (2)
Pain - Grade 2 (General disorders) | 0 (0) | 2 (3)
Pain - Grade 3 (General disorders) | 0 (0) | 1 (1)
Pyrexia - Grade 1 (General disorders) | 0 (0) | 2 (2)
Temperature intolerance - Grade 1 (General disorders) | 0 (0) | 1 (1)
Tenderness - Grade 1 (General disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia - Grade 1 (Hepatobiliary disorders) | 0 (0) | 1 (2)
Hyperbilirubinaemia - Grade 2 (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity - Grade 2 (Immune system disorders) | 0 (0) | 1 (1)
Candidiasis - Grade 1 (Infections and infestations) | 1 (1) | 0 (0)
Ear infection - Grade 1 (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection - Grade 1 (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex - Grade 1 (Infections and infestations) | 1 (1) | 0 (0)
Influenza - Grade 1 (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis - Grade 1 (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis - Grade 2 (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis - Grade 1 (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia - Grade 2 (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis - Grade 1 (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection - Grade 1 (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection - Grade 2 (Infections and infestations) | 2 (2) | 1 (1)
Sunburn - Grade 1 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn - Grade 1 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged - Grade 1 (Investigations) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged - Grade 2 (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased - Grade 1 (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased - Grade 1 (Investigations) | 0 (0) | 2 (2)
Blood albumin decreased - Grade 1 (Investigations) | 0 (0) | 2 (2)
Blood bicarbonate decreased - Grade 1 (Investigations) | 0 (0) | 1 (1)
Blood chloride increased - Grade 1 (Investigations) | 0 (0) | 2 (2)
Blood creatine increased - Grade 1 (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased - Grade 1 (Investigations) | 0 (0) | 2 (2)
Blood creatinine increased - Grade 2 (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased - Grade 3 (Investigations) | 0 (0) | 1 (1)
Blood phosphorus - Grade 1 (Investigations) | 0 (0) | 1 (1)
Blood potassium increased - Grade 1 (Investigations) | 0 (0) | 1 (1)
Blood urea increased - Grade 1 (Investigations) | 0 (0) | 1 (1)
Blood uric acid increased - Grade 1 (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased - Grade 2 (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased - Grade 3 (Investigations) | 1 (2) | 0 (0)
Hepatic enzyme increased - Grade 1 (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased - Grade 2 (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal - Grade 2 (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased - Grade 2 (Investigations) | 0 (0) | 2 (3)
Neutrophil count decreased - Grade 4 (Investigations) | 0 (0) | 2 (2)
Platelet count decreased - Grade 2 (Investigations) | 0 (0) | 1 (1)
Platelet count decreased - Grade 3 (Investigations) | 0 (0) | 3 (3)
Protein total decreased - Grade 1 (Investigations) | 0 (0) | 3 (3)
Protein total decreased - Grade 2 (Investigations) | 0 (0) | 1 (1)
Prothrombin level abnormal - Grade 1 (Investigations) | 0 (0) | 1 (1)
Weight decreased - Grade 1 (Investigations) | 0 (0) | 1 (1)
Weight decreased - Grade 2 (Investigations) | 0 (0) | 1 (1)
Weight increased - Grade 1 (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased - Grade 2 (Investigations) | 0 (0) | 1 (1)
Anorexia - Grade 1 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite - Grade 1 (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
Decreased appetite - Grade 2 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration - Grade 1 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid retention - Grade 1 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia - Grade 1 (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Hyperglycaemia - Grade 3 (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia - Grade 1 (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hyperkalaemia - Grade 2 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypermagnesaemia - Grade 1 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperphosphataemia - Grade 1 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperphosphataemia - Grade 2 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricaemia - Grade 1 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia - Grade 1 (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hypoalbuminaemia - Grade 2 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia - Grade 1 (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hypocalcaemia - Grade 2 (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypocalcaemia - Grade 3 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia - Grade 1 (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalaemia - Grade 1 (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalaemia - Grade 2 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia - Grade 1 (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia - Grade 3 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoproteinaemia - Grade 1 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia - Grade 1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Arthralgia - Grade 2 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Back pain - Grade 2 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Flank pain - Grade 2 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms - Grade 1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal discomfort - Grade 1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in jaw - Grade 1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumour flare - Grade 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (5)
Tumour flare - Grade 2 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amnesia - Grade 1 (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion - Grade 2 (Nervous system disorders) | 0 (0) | 1 (1)
Disturbance in attention - Grade 1 (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness - Grade 1 (Nervous system disorders) | 2 (3) | 7 (8)
Dizziness - Grade 2 (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness - Grade 3 (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness postural - Grade 1 (Nervous system disorders) | 0 (0) | 1 (1)
Headache - Grade 1 (Nervous system disorders) | 0 (0) | 3 (3)
Headache - Grade 2 (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia - Grade 1 (Nervous system disorders) | 1 (1) | 2 (4)
Hypoaesthesia - Grade 2 (Nervous system disorders) | 0 (0) | 1 (2)
Memory impairment - Grade 1 (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy - Grade 1 (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral - Grade 1 (Nervous system disorders) | 0 (0) | 5 (6)
Paraesthesia - Grade 1 (Nervous system disorders) | 2 (3) | 0 (0)
Sinus headache - Grade 1 (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence - Grade 1 (Nervous system disorders) | 0 (0) | 1 (1)
Tremor - Grade 1 (Nervous system disorders) | 1 (2) | 5 (6)
Anxiety - Grade 1 (Psychiatric disorders) | 0 (0) | 2 (2)
Confusional state - Grade 1 (Psychiatric disorders) | 0 (0) | 2 (2)
Depression - Grade 1 (Psychiatric disorders) | 0 (0) | 2 (2)
Depression - Grade 2 (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia - Grade 1 (Psychiatric disorders) | 1 (1) | 2 (2)
Insomnia - Grade 2 (Psychiatric disorders) | 0 (0) | 1 (1)
Mood swings - Grade 1 (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure - Grade 2 (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention - Grade 1 (Renal and urinary disorders) | 0 (0) | 1 (1)
Asthma - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dysphonia - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Dyspnoea - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Dyspnoea exertional - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Nasal congestion - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry skin - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Erythema - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypoaesthesia facial - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail disorder - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats - Grade 2 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (6)
Pruritus - Grade 2 (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus generalised - Grade 2 (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash - Grade 1 (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (7)
Rash - Grade 2 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash generalised - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
Rash generalised - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash generalised - Grade 3 (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Rash pruritic - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash pruritic - Grade 3 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin exfoliation - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin odour abnormal - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension - Grade 1 (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was stopped early due to low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No